CLINICAL TRIAL: NCT02776254
Title: Community ART for Retention in Zambia: Evaluating the Feasibility, Effectiveness, and Efficiency of Decentralized and Streamlined Antiretroviral Therapy Care Models
Brief Title: Differentiated Care for Improved Health Systems Efficiency and Health Outcomes in Zambia
Acronym: CommART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Johns Hopkins University (Other); University of Alabama at Birmingham (Other); University of California, San Francisco (Other); American Institutes for Research (Other); University of Zambia (Other); Ministry of Health, Zambia (Other Government); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ID OPP1105306
Record Dates: First submitted 2016-03-13; First posted 2016-05-18 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: HIV
Keywords: anti-retroviral therapy; differentiated care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- START (Experimental): The START model aims to deliver a higher intensity of treatment services by offering same-day CD4 testing and results, streamlined adherence counseling, and quicker initiation of life-long ART to patients enrolling in HIV care and treatment services.
  Interventions: Other: START
- FAST Track (Experimental): In the FAST-TRACK model a pharmacy technician will dispense drugs) and lay health care workers will provide brief symptom screening to identify patients in need of higher-level care. If there is no need of higher-level care, then the clinic visit is over.
  Interventions: Other: FAST-TRACK
- CAG (intervention) (Experimental): CAG intervention, consists of facilitated groups of six people based on geographic proximity of home address and patient preference. This group of six people, will meet monthly at a designated place in the community to provide support and receive medications. Each month one of the members will rotate visiting the clinic for their routine medical visit and will pick up medications for the entire CAG and bring them back to the community. This rotation schedule will recur every six months. Lay health care workers will provide brief symptom screening to identify patients in the group that need of higher-level care.
  Interventions: Other: CAG
- CAG (comparison) (Active Comparator): Eligible patients at control sites will be approached for willingness to participate in the study. Those who are willing will be enrolled in the study and consent will be obtained to use patient data within SmartCare to evaluate the primary outcome of retention.
  Interventions: Other: CAG
- UAG (intervention) (Experimental): Urban sites will be eligible for the UAG model in which patients will be joined into a UAG group consisting of 30 people. Each UAG group will meet every two to three months at a designated site (either at the clinic facility or another site in the community). Patients will receive (a) group adherence counseling led by a lay HCW (b) two to three month supply of ART medications via a pharmacy tech (c) attendance record and symptom assessment. As in the CAG model, patients may be referred up-referred for care based on acute illness or patient preference. Patients will continue to visit the facility for a routine medical visit with a professional HCW every six months.
  Interventions: Other: UAG
- UAG (comparison) (Active Comparator): Eligible patients at control sites will be approached for willingness to participate in the study. Those who are willing will be enrolled in the study and consent will be obtained to use patient data within SmartCare to evaluate the primary outcome of retention.
  Interventions: Other: UAG

INTERVENTIONS:
Other: START — Point of care testing for rapid ART initiation
  Arms: START
Other: CAG — Community Adherence Group
  Arms: CAG (comparison); CAG (intervention)
Other: UAG — Urban Adherence Group
  Arms: UAG (comparison); UAG (intervention)
Other: FAST-TRACK — Prescription refill only
  Arms: FAST Track

SUMMARY:
This study seeks to create generalizable knowledge about the implementation process as well as the effectiveness and efficiency of a differentiated care system, by measuring patient health outcomes and implementation outcomes such as acceptability, feasibility, fidelity, and costs

DETAILED DESCRIPTION:
This is a joint endeavor of the Zambian Ministry of Health (MoH), Ministry of Community Development, Mother & Child Health (MCDMCH) and the Centre for Infectious Disease Research in Zambia (CIDRZ) with funding from the Bill & Melinda Gates Foundation.

The study evaluates four models of streamlined HIV care in reducing patients' time and cost: (1) community adherence groups (CAG), (2) urban adherence groups (UAG), (3) Fast-Track clinic visits and (4) streamlined ART initiation (START). CAG and UAG are assessed using a cluster-randomized design; Fast-Track and START using an observational approach to compare changes in the outcome through a difference in difference approach.

1. Specific Objectives

Objective 1:

To determine acceptability, appropriateness, and feasibility of a differentiated care system in Zambia, by assessing perspectives of (1) patients and family members (2) health care workers and (3) government and local leaders.

Objective 2:

To evaluate effectiveness (retention), efficiency (cost-effectiveness), and health care quality (quantitative and qualitative measures) of a differentiated and targeted care system.

Objective 3:

To develop a "methodologic" toolkit for assessment of local needs, preferences and scale-up of differentiated care models in varied contexts, using data from Objectives 1 and 2.

2.0 Methodology 2.1 Objective 1 Mixed methods approach will be used to evaluate perceptions on challenges in accessing and adhering to life-long HIV treatment and to assess needs/preferences for differentiated care models collected from patients and family members (demand side), health facilities -professional and community health workers (supply side), and government and local leaders using in-depth interviews (IDIs), focus group discussions (FGDs), and discrete choice surveys (DCS) to sequentially analyze supply and demand side factors that may influence uptake.

Population Key government and other stakeholders in HIV or other relevant community based service delivery will be interviewed. Professional and lay health workers in ART program, Pre-ART and ART patients and, a sample of household members of ART or pre-ART patient registered at selected health facility will be interviewed.

Measurements/Procedures For Objective 1: IDIs, FGDs, medical chart reviews, DCS/general survey Semi-structured guides by participant type will be used to conduct IDIs and FGDs in English or a local language (Nyanja, Bemba, or Tonga). Where permitted, IDIs/FGDs will be audio-recorded for transcription and analysis. Participants will be reimbursed for travel. IDIs will last 1 and FGDs 1-2 hours.

A cross-sectional survey will be used to measure patient access and psychosocial needs. Access needs will be assessed by questions on appropriateness of current clinic operating hours; distance, cost, and time to reach clinic; household income, assets, and expenditures; and opportunity costs of a clinic visit. Patient costs related to health care utilization, including transport, communication, and food costs will be elicited. To assess psychosocial needs, validated scales and indices to measure stigma (Revised Berger), depression (PHQ-9), alcohol consumption (AUDIT-C), and domestic violence will be applied. The survey administered in the language of participant's choice by trained survey enumerators using tablets will take approximately 30-45 minutes and uploaded to the central database.

The electronic clinical information system (SmartCare) will be utilized to evaluate patient clinical needs. Distribution of clinical needs will be assessed for degree of immunosuppression at entry into care, frequency of opportunistic infections after treatment initiation, and frequency of "ill" versus "healthy" visits.

DCSs will be used to assess patient preference for different, discrete characteristics of various models of community-based ART delivery. All possible combinations of key attributes/aspects of community-based ART models and number of levels/options for them will be put in subsets divided in blocks. Each participant is asked only one possible block of about 10 questions.

Analytic Approach Qualitative data will be imported into software for managing qualitative analysis (e.g. N-Vivo or Atlas TI), iteratively coded and cross-referenced with survey data. Scale scores may be analyzed using descriptive statistics and linear regression modeling. For DCS, main effects plus two-way interactions between different parameters will be estimated using a nested logit framework.

Sampling Approach/Sample Size Considerations The convenience sample consists of 20 IDIs with government and community leaders; two FGDs each with professional HCW, Lay HCW and family members from1 urban and 1 rural clinic in each province; 4 FGDs with ART patients (2 urban and 2 rural clinic) in each province; and 2 FGDs with pre-ART patients (1 urban and 1 rural clinic) in Lusaka province only.

General survey: 1,600 patients (of which 800 are ART and 800 are pre-ART). A precision approach was used to calculate number of ART and pre-ART participants respectively necessary to estimate a binary indicator with 5% margin of error and 95% confidence interval, assuming a prevalence of p=0.5 and a design effect of 2 [ n=((1.96^2) * 0.5* 0.5 *2)/(0.05^2)=768].

2.2 Objective 2: To evaluate the effectiveness, efficiency, and health care quality of a differentiated system of care that includes targeted models of care.

Effectiveness of a differentiated system of HIV care delivery in which frequency, type, or intensity of contact with the health system is tailored to patient needs will be evaluated. CAGs, UAGs, fast-track, and START will be simultaneously implemented and evaluated using a common evaluation framework that includes effectiveness (retention), efficiency, and quality.

Methodology A matched cluster randomized design approach is proposed for CAG and UAG models to account for the clinic-level intervention and possible selection bias. With little to no observational/ implementation data for Fast-Track and START models globally, a difference-in-difference design will be used to calculate effect of the models on outcomes.

Population See inclusion and exclusion criteria Procedures Description of Interventions: Entered elsewhere

Patient recruitment:

At all intervention sites: Facility staff will identify eligible patients during routine clinic visits and notify the study research assistant about potential study participants. The research study assistant will assess patient willingness to participate in the intervention and will obtain informed consent for study participation.

START model: Staff will use national guidelines to determine ART eligibility and, with participants' informed consent, expedite provision of on-site CD4 testing using point of care platform for all newly diagnosed and ART-naive patients due for routine CD4 monitoring. Participants will not be actively followed in the 12-months after ART initiation.

At control sites: Eligible patients at control sites, willing to join CAG and UAG studies, will be enrolled. Consent will be obtained to extract their SmartCare data.

Baseline viral load testing:

For participants enrolled into CAG, UAG and Fast-Track intervention, dry blood spot specimens will be obtained via finger prick. Specimens will be transmitted to CIDRZ central laboratory for baseline viral load testing. Results will be communicated to providers and patients and, documented in SmartCare.

Costing A subset of participants in each model will be interviewed on direct and indirect health costs of the intervention using a semi-structured questionnaire. Administrative data may also be used.

Exit viral load testing and patient exit-survey All participants will have an exit viral load test in the 12th month. In CAG, UAG, and Fast-Track models, a patient exit-survey will assess patient satisfaction and patient centeredness.

Measurements Standard de-identified socio-demographic, laboratory and clinical data will be extracted from SmartCare.

Information in model-specific registers (attendance, receipt of medications, symptom checklist, patient preference between intervention and standard care, up-referral due to presence of symptoms or a patient's desire to return to standard care, or down-referral to model when patients with acute illness stabilize) will be entered into the study database using a tablet.

Patient satisfaction and centeredness will be captured by the semi-structured patient-exit survey conducted after the 12-month intervention period.

Baseline and exit viral load testing will be conducted. A semi-structured costing questionnaire used with a subset of intervention participants will assess related direct and indirect health costs. To calculate resource use of each activity, time-in-motion studies will be conducted among patients and health care workers prior to and during the intervention.

Process data will be collected facility-level assessments of pharmacy stock outs and through HCW interviews at end of follow-up period.

Analytic Approach For START, date of ART initiation is the primary outcome. For CAG and UAG interventions, Kaplan-Meier estimates of time to the primary outcome, stratified by intervention condition, using log rank tests will be calculated. For Fast-track and START, primary analysis will take a difference-in-difference approach to estimate difference in the change in the rate of the outcome in intervention settings. In secondary analyses of the primary outcome, longer intervals of lateness that comprise a missed pharmacy visit (14 and 30 days) as well as adjustment for baseline patient characteristics will be explored along with analysis using medication possession ratio (MPR) as the outcome and other metrics of retention that incorporate both frequency of missed visit and interval of time before return.

Sample Size Considerations CAG/UAG: Program data suggest that 65% of patients are > 7 days late for a pharmacy refill visit in their first year of ART in 95% (+15%) of clinics. Assuming a conservative matched co-efficient of variation of 0.10 and a 50% reduction in missed pharmacy visits, selection of five clinics and 90 patients per site will yield power of 96% for CAG intervention. Under more conservative assumptions about between clinic variability and the effect size, this sample size yields >80% power. For UAG intervention, target sample size is 4 UAGs of 30 people each in five intervention sites (120 participants per site; 600 across sites). Under the same assumptions as the CAG model, this sample size yields power of > 90% and is robust to varying assumptions about correlation.

Fast-track: Targeting 200 patients at each of four sites (2 intervention and 2 control sites), a fall to 40% of the assumed 80% patients that miss a pharmacy visit in the first year, gives 80% power.

START: Assuming ART initiation at 2 weeks rises from 60% to 85%, 100 patients at each of eight sites (4 intervention and 4 control sites; n=800), rho of 0.15 yields an anticipated power of 78%.

2.3 Objective 3: Methodological Toolkit After data synthesis, a methodological toolkit will be developed to guide assessment of feasibility, acceptability, needs, preferences and implementation for differentiated care models. Data will be collected using work process tracking and costing; and interviews with study staff and key decision makers. The toolkit will be easily digestible and lead to actionable plans to move from current to differentiated care models in differing circumstances and contexts. With input from reviewers, the toolkit will be finalized and digital and hard copies will be distributed at dissemination events with the MoH, MCDMCH and other national and sub-national stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive adolescents and adults (> 14 years of age)
* Last CD4 count (obtained within the last six months) > 200
* Not acutely ill
* For CAGs, UAGs, and Fast-Track models: on ART for at least 6 months
* For the START model: ART naïve and meet the Zambian HIV guidelines for treatment initiation

Exclusion Criteria:

* For CAGs, UAGs: Inability to participate in the group activities due to cognition deficits or mental illness.
* Unable to provide consent or unwilling to participate in study
* Pregnancy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Retention in care (Time to first missed pharmacy pick-up) | 12 months
  Time to first missed pharmacy pick-up (>7 days)

SECONDARY OUTCOMES:
Feasibility of implementing differentiated care from stakeholder perspectives | 12 months
  stakeholders' perceptions on factors that facilitate or impede delivery of differential models of care through qualitative assessments (i.e. HCW interviews at end of follow-up period).
Feasibility of implementing differentiated care based on ART availability | 12 months
  facility-level assessments (i.e. frequency of pharmacy stock outs) that facilitate or impede delivery of differential models of care
Activity Based Costing (cost per activity based on Time and Motion) | 12 months
  Cost per activity will be estimated using time-in-motion forms among health care workers prior to and during implementation
Cost to patient based on semi-structured interviews | 12 months
  Cost will be estimated through a semi-structured costing questionnaire administered to a subset of intervention participants to assess direct and indirect health costs of the intervention.
Research Costs (cost of conducting implementation science) | 12 months
  Activity-based cost of researching differentiated care based on budgets and spending reports
Fidelity by monitoring the proportion of eligible patients successfully enrolled and retained in a model. | 12 months
  proportion of eligible patients successfully enrolled and retained in a model
Access to care (time in days from positive symptom screen to appropriate referral) | 12 months
  Time (days) from positive symptom screen to appropriate referral
Efficiency (Difference between cost per additional patient retained and the cost per death averted divided by the difference in their effect) | 12 months
  Difference between Incremental cost per additional patient retained and the cost per death averted divided by the difference in their effect
Proportion of patients with appropriate laboratory monitoring (CD4 count testing) | every 6 months for a year
  As this is an assessment of models of delivering ART in a manner more efficient than presentation to clinician every month, safety is estimated by appropriate referral based on laboratory monitoring by clinical staff (CD4 count every 6 months for a year)
Proportion of patients with appropriate laboratory monitoring through viral load testing | 12 months
  As this is an assessment of models of delivering ART in a manner more efficient than presentation to clinician every month, safety is estimated by appropriate referral based on laboratory monitoring by clinical staff (Viral load every 12 months)
Proportion of patients with appropriate symptom screening | Every 1-3 months for 12 months
  As this is an assessment of models of delivering ART in a manner more efficient than presentation to clinician every month, safety is estimated by appropriate referral based on symptom screening by study staff (every 1-3 months per year)
Retention rate disaggregated by age (adult and adolescent) | 12 months
  Comparison of retention rates between adults and adolescents will be used as a measure of equity
Retention rate disaggregated by sex (male and female) | 12 months
  Comparison of retention rates between men and women will be used as a measure of equity
Proportion of patients virally suppressed at one year among those exposed to the intervention compared to control conditions using mixed effects logistic regression | 12 months
  Viral suppression should be comparable between the intervention and control groups to ascertain whether patient outcomes are better or at least the same as current routine practice
Patient satisfaction using patient exit-survey | 12 months
  Effect of the intervention on patient satisfaction through mixed effects linear regression

CONTACTS AND LOCATIONS:
Overall Officials: Charles Holmes, MD, MPH, Principal Investigator — Centre for Infectious Disease Research in Zambia; Izukanji Sikazwe, MBChB, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Health ZMo. UNAIDS Country Progress Report Zambia. March 31, 2012 2012.
- [Background] Humphreys CP, Wright J, Walley J, Mamvura CT, Bailey KA, Ntshalintshali SN, West RM, Philip A. Nurse led, primary care based antiretroviral treatment versus hospital care: a controlled prospective study in Swaziland. BMC Health Serv Res. 2010 Aug 5;10:229. doi: 10.1186/1472-6963-10-229. PMID 20687955
- [Background] Kipp W, Konde-Lule J, Saunders LD, Alibhai A, Houston S, Rubaale T, Senthilselvan A, Okech-Ojony J. Antiretroviral treatment for HIV in rural Uganda: two-year treatment outcomes of a prospective health centre/community-based and hospital-based cohort. PLoS One. 2012;7(7):e40902. doi: 10.1371/journal.pone.0040902. Epub 2012 Jul 17. PMID 22815862
- [Background] Jaffar S, Amuron B, Foster S, Birungi J, Levin J, Namara G, Nabiryo C, Ndembi N, Kyomuhangi R, Opio A, Bunnell R, Tappero JW, Mermin J, Coutinho A, Grosskurth H; Jinja trial team. Rates of virological failure in patients treated in a home-based versus a facility-based HIV-care model in Jinja, southeast Uganda: a cluster-randomised equivalence trial. Lancet. 2009 Dec 19;374(9707):2080-2089. doi: 10.1016/S0140-6736(09)61674-3. Epub 2009 Nov 24. PMID 19939445
- [Background] Kredo T, Ford N, Adeniyi FB, Garner P. Decentralising HIV treatment in lower- and middle-income countries. Cochrane Database Syst Rev. 2013 Jun 27;2013(6):CD009987. doi: 10.1002/14651858.CD009987.pub2. PMID 23807693
- [Background] Luque-Fernandez MA, Van Cutsem G, Goemaere E, Hilderbrand K, Schomaker M, Mantangana N, Mathee S, Dubula V, Ford N, Hernan MA, Boulle A. Effectiveness of patient adherence groups as a model of care for stable patients on antiretroviral therapy in Khayelitsha, Cape Town, South Africa. PLoS One. 2013;8(2):e56088. doi: 10.1371/journal.pone.0056088. Epub 2013 Feb 13. PMID 23418518
- [Background] Decroo T, Koole O, Remartinez D, dos Santos N, Dezembro S, Jofrisse M, Rasschaert F, Biot M, Laga M. Four-year retention and risk factors for attrition among members of community ART groups in Tete, Mozambique. Trop Med Int Health. 2014 May;19(5):514-21. doi: 10.1111/tmi.12278. Epub 2014 Feb 12. PMID 24898272
- [Background] Decroo T, Telfer B, Biot M, Maikere J, Dezembro S, Cumba LI, das Dores C, Chu K, Ford N. Distribution of antiretroviral treatment through self-forming groups of patients in Tete Province, Mozambique. J Acquir Immune Defic Syndr. 2011 Feb 1;56(2):e39-44. doi: 10.1097/QAI.0b013e3182055138. PMID 21084990
- [Background] Fairall L, Bachmann MO, Lombard C, Timmerman V, Uebel K, Zwarenstein M, Boulle A, Georgeu D, Colvin CJ, Lewin S, Faris G, Cornick R, Draper B, Tshabalala M, Kotze E, van Vuuren C, Steyn D, Chapman R, Bateman E. Task shifting of antiretroviral treatment from doctors to primary-care nurses in South Africa (STRETCH): a pragmatic, parallel, cluster-randomised trial. Lancet. 2012 Sep 8;380(9845):889-98. doi: 10.1016/S0140-6736(12)60730-2. Epub 2012 Aug 15. PMID 22901955
- [Background] Brennan AT, Long L, Maskew M, Sanne I, Jaffray I, MacPhail P, Fox MP. Outcomes of stable HIV-positive patients down-referred from a doctor-managed antiretroviral therapy clinic to a nurse-managed primary health clinic for monitoring and treatment. AIDS. 2011 Oct 23;25(16):2027-36. doi: 10.1097/QAD.0b013e32834b6480. PMID 21997488
- [Background] Babigumira JB, Castelnuovo B, Stergachis A, Kiragga A, Shaefer P, Lamorde M, Kambugu A, Muwanga A, Garrison LP. Cost effectiveness of a pharmacy-only refill program in a large urban HIV/AIDS clinic in Uganda. PLoS One. 2011 Mar 28;6(3):e18193. doi: 10.1371/journal.pone.0018193. PMID 21464895
- [Background] Selke HM, Kimaiyo S, Sidle JE, Vedanthan R, Tierney WM, Shen C, Denski CD, Katschke AR, Wools-Kaloustian K. Task-shifting of antiretroviral delivery from health care workers to persons living with HIV/AIDS: clinical outcomes of a community-based program in Kenya. J Acquir Immune Defic Syndr. 2010 Dec;55(4):483-90. doi: 10.1097/QAI.0b013e3181eb5edb. PMID 20683336
- [Background] Bemelmans M, Baert S, Goemaere E, Wilkinson L, Vandendyck M, van Cutsem G, Silva C, Perry S, Szumilin E, Gerstenhaber R, Kalenga L, Biot M, Ford N. Community-supported models of care for people on HIV treatment in sub-Saharan Africa. Trop Med Int Health. 2014 Aug;19(8):968-77. doi: 10.1111/tmi.12332. Epub 2014 May 28. PMID 24889337
- [Background] Rosen S, Fox MP. Retention in HIV care between testing and treatment in sub-Saharan Africa: a systematic review. PLoS Med. 2011 Jul;8(7):e1001056. doi: 10.1371/journal.pmed.1001056. Epub 2011 Jul 19. PMID 21811403
- [Background] Rasschaert F, Telfer B, Lessitala F, Decroo T, Remartinez D, Biot M, Candrinho B, Mbofana F, Van Damme W. A qualitative assessment of a community antiretroviral therapy group model in Tete, Mozambique. PLoS One. 2014 Mar 20;9(3):e91544. doi: 10.1371/journal.pone.0091544. eCollection 2014. PMID 24651523
- [Background] Hickey MD, Salmen CR, Omollo D, Mattah B, Fiorella KJ, Geng EH, Bacchetti P, Blat C, Ouma GB, Zoughbie D, Tessler RA, Salmen MR, Campbell H, Gandhi M, Shade S, Njoroge B, Bukusi EA, Cohen CR. Implementation and Operational Research: Pulling the Network Together: Quasiexperimental Trial of a Patient-Defined Support Network Intervention for Promoting Engagement in HIV Care and Medication Adherence on Mfangano Island, Kenya. J Acquir Immune Defic Syndr. 2015 Aug 1;69(4):e127-34. doi: 10.1097/QAI.0000000000000664. PMID 25984711
- [Derived] Bolton Moore C, Pry JM, Mukumbwa-Mwenechanya M, Eshun-Wilson I, Topp S, Mwamba C, Roy M, Sohn H, Dowdy DW, Padian N, Holmes CB, Geng EH, Sikazwe I. A controlled study to assess the effects of a Fast Track (FT) service delivery model among stable HIV patients in Lusaka Zambia. PLOS Glob Public Health. 2022 Aug 3;2(8):e0000108. doi: 10.1371/journal.pgph.0000108. eCollection 2022. PMID 36962510
- [Derived] Roy M, Bolton-Moore C, Sikazwe I, Mukumbwa-Mwenechanya M, Efronson E, Mwamba C, Somwe P, Kalunkumya E, Lumpa M, Sharma A, Pry J, Mutale W, Ehrenkranz P, Glidden DV, Padian N, Topp S, Geng E, Holmes CB. Participation in adherence clubs and on-time drug pickup among HIV-infected adults in Zambia: A matched-pair cluster randomized trial. PLoS Med. 2020 Jul 1;17(7):e1003116. doi: 10.1371/journal.pmed.1003116. eCollection 2020 Jul. PMID 32609756
- [Derived] Tucker A, Tembo T, Tampi RP, Mutale J, Mukumba-Mwenechanya M, Sharma A, Dowdy DW, Moore CB, Geng E, Holmes CB, Sikazwe I, Sohn H. Redefining and revisiting cost estimates of routine ART care in Zambia: an analysis of ten clinics. J Int AIDS Soc. 2020 Feb;23(2):e25431. doi: 10.1002/jia2.25431. PMID 32064766
- See also: Frontieres MS. Community ART Group Toolkit: How to Implement the CAG Model. http://www.msf.org/sites/msf.org/files/cag_toolkit.pdf. Accessed August 28, 2014 — http://www.msf.org/sites/msf.org/files/cag_toolkit.pdf